CLINICAL TRIAL: NCT05382520
Title: Sensory Rehabilitation in Chemotherapy Induced Peripheral Neuropathy (CIPN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Zefat Academic College (Other)
Responsible Party: Principal Investigator, Rotem Merose, Breast Oncologist, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0057-22-ASF
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: CIPN
Keywords: Neuropathic pain; Chemo Induced Peripheral Neuropathy (CIPN); Sensory rehabilitation; Explicit Sensory Retraining
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Prospective Pilot and Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Explicit sensory retraining for lower extremity in individuals with CIPN (Experimental): Explicit sensory retraining for lower extremity function (pain, sensory, balance, gait). five one-hour sessions, a week apart: Pre-Post assessment sessions with 3 treatment sessions in between. Home exercise assigned.
  Interventions: Diagnostic Test: Questionares and practice

INTERVENTIONS:
Diagnostic Test: Questionares and practice — Questionares and practice

SUMMARY:
Physiotherapist research about Sensory rehabilitation in chemotherapy induced peripheral neuropathy (CIPN) with the aid of questioners and physiotherapy practice

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over who suffer from chemotherapy-induced neuropathy (CIPN), according to the patient's report, more than 3 months since the end of the chemotherapy treatment.

Exclusion Criteria:

1. Sensory damage / neuropathy that existed even before the start of chemotherapy
2. Incidents of recurrent falls even before the start of chemotherapy (over 2 falls for 6 months)
3. Central nervous system involvement
4. Major pre-morbid orthopedic lower limb impairment
5. Hebrew language not sufficient for assessment and treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
TNAS | 2 years
  TNAS -Treatment-Induced Neuropathy Assessment Scale. 0-90. higher score = worse status
VAS | 2 years
  0-100 mm visual scale: self-reporting pain assessment from no pain to worst pain possible. We will ask for current pain and the worst pain during the last week.
FABS | 2 years
  Fullerton Advanced Balance Scale: high function balance test - consisting of 10 activities in both static and dynamic phases; 10-40, higher scores are better.
TUG | 2 years
  Timed Up and Go: fall prediction screening test; measures time taken to raise from a chair walking 3 meters and re-sit.
NSA | 2 years
  Nottingham Sensory Assessment: sensory detection and discrimination test
Semmes-Weinstein monofilament testing | 2 years
  tactile detection threshold
LEPT | 2 years
  Lower Extremity Position Test: proprioception detection and quantification
Allodynia | 2 years
  tested by non-painful mechanical stimulation: gentle brushing and monofilament

CONTACTS AND LOCATIONS:
Overall Officials: Rotem Merose, Dr., Principal Investigator — Assaf Harofee MC
Locations (1):
- Shamir medical center, Beer Yaaqov, Israel

IPD SHARING:
Plan to Share IPD: Undecided